CLINICAL TRIAL: NCT05784519
Title: Clinical Study of Mesenchymal Stem Cell Eye Drops for Treating Dry Eye Disease
Brief Title: Therapeutic Effect of Stem Cell Eye Drops on Dry Eye Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC202200102
Record Dates: First submitted 2023-02-21; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-12

CONDITIONS: Mesenchymal Stem Cell; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): The MSCs eye drops was administered to enrolled patients with 5×10^5 /50μl in each eye, twice a day for 2 weeks.
  Interventions: Drug: MSCs eye drops

INTERVENTIONS:
Drug: MSCs eye drops — MSCs were used to prepare single-cell suspension, and 0.9% sodium chloride was added to balance PH value to prepare the effective, safe and stable eye drops. Giving the patient with 5×10^5 /50μl in each eye, twice a day for 2 weeks.

SUMMARY:
The goal of this non-randomized, prospective, open, one-arm clinical study is to learn about the clinical efficacy of stem cell eye drops in patients with dry eye disease (DED) who failed to respond to artificial tear sodium hyaluronate eye drops three times a day for two weeks.

The main question aims to answer are:

* How effective are stem cell eye drops in patients with DED?
* How safe are stem cell eye drops for patients with DED? Participants will be treated with mesenchymal stem cells (MSCs) eye drops, 5×10^5 /50μl in each eye, twice a day for two weeks and they will be followed up for three months after treatment.

DETAILED DESCRIPTION:
This study was mainly divided into three parts: screening period, treatment period and late treatment period. (1) Screening period: For the DED patients with artificial tear sodium hyaluronate drops three times a day and no effect for two consecutive weeks, OSDI score, fluorescein sodium stain score, tear secretion test and tear film rupture time examination were performed. 10 eligible subjects were screened out according to the inclusion/exclusion criteria, and the subjects were asked to sign informed consent. Relevant clinical examination data were collected and subjects were enrolled. 1) OSDI questionnaire: it was divided into 3 dimensions, including ocular symptoms, visual function, and environmental factors.2) Fluorescein staining score of ocular surface: After staining with 0.25% fluorescein sodium, defect staining was observed under slit lamp microscope. Cornea was scored in 3 areas: top, center and bottom. Each area was scored by 0 points (without any staining), 1 points (partial staining), 2 points (staining of more than half of the area), and 3 points (staining of the whole area). The total was divided into the sum of 3 areas. A higher score indicates more severe ocular surface damage. 3) Schirmer test: Standard tear test paper was taken and held in the conjunctival sac at 1/3 of the lower outer eyelid, and the patient was instructed to close the eyes gently. The results were observed 5 minutes later. The tear secretion test < 10mm/5min was abnormal. 4) Tear break-up time: After staining with 0.25% fluorescein sodium, patients were instructed to close their eyes under the slit lamp microscope. The tear film rupture time was calculated from the time of eye opening to the appearance of the first burst spot, and the average value was taken for three consecutive tests. The rupture time of tear film was less than 10s. (2) Treatment period: Formal clinical treatment: 10 enrolled patients received MSC eye drops twice a day for two weeks. OSDI score, ocular fluorescein sodium stain score, tear secretion test and tear film rupture time examination were performed every weekend during drug administration. Adverse events, serious adverse events and drug-related adverse events ≥Ⅲ during treatment were recorded to evaluate drug safety. (3) Late treatment: 3 months of follow-up after the end of treatment. OSDI score was performed during weekly telephone follow-up, and clinical indicators (OSDI score, fluorescein sodium staining score of ocular surface, tear secretion test and tear film rupture time test) were examined every four weeks to evaluate the treatment effect of DED.

ELIGIBILITY:
1. Inclusion Criteria:

   1. As determined by the investigator, the subject is able to understand and comply with the protocol requirements;
   2. Subject or subject's legal representative (if applicable) sign and date the written informed consent or any privacy authorization document required prior to the commencement of the study process;
   3. Age 40-60;
   4. Female patients;
   5. The subject has received artificial tear sodium hyaluronate treatment with eye drops three times a day, but the treatment has no effect for two weeks, and the clinical examination results are consistent with:

      * OSDI score ≥13;
      * Schirmer test < 10mm/5min;
      * Tear break-up time < 10s;
      * Fluorescein sodium staining on the ocular surface was positive.
2. Exclusion Criteria:

   1. Eye exclusion criteria:

      * Subjects with other eye diseases such as glaucoma, cataract, uveitis, optic neuritis, etc.；
      * The subjects had undergone eye surgery (e.g., cataract surgery) within the last three months;
      * Subjects who wear contact lenses for a long time and are unwilling to remove them in the study;
      * The subject has received eye drops in the past 24 hours that may affect the clinical study.
   2. Exclusion criteria related to infectious diseases:

      * The subject has fungal, bacterial or viral keratitis or conjunctivitis with evidence of infection;
      * The subject has chronic hepatitis B virus (HBV) infection or chronic hepatitis C virus (HCV) infection;
      * The subject has any identified congenital or acquired immunodeficiency (e.g., common immunodeficiency, human immunodeficiency HIV infection, organ transplantation);
      * The subject has active tuberculosis (TB positive);
      * Subjects receive any live vaccine within 30 days prior to screening.
   3. Exclusion criteria for general circumstances:

      * The subject is allergic to the stem cell eye drops;
      * The subject has any unstable or uncontrolled cardiovascular, pulmonary, liver, kidney, gastrointestinal, urogenital, hematological, clotting, immunological, endocrine/metabolic, or other medical condition that the investigator deems to interfere with the study or endanger the safety of the subject;
      * Subjects had had any surgery requiring general anesthesia within 30 days prior to enrollment, or planned to have a larger procedure during the study period surgery;
      * Subjects have a history of severe neurological diseases, including stroke, multiple sclerosis, brain tumors, or neurodegenerative diseases；
      * The subjects had active psychosis, which the researchers thought might interfere with their compliance with the study process;
      * Lactating female subjects, or female subjects with positive serum pregnancy test results during the screening period, or positive urine pregnancy test results prior to study drug administration.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The change of OSDI score | 1 week
  OSDI questionnaire: It was divided into 3 dimensions, including ocular symptoms, visual function, and environmental factors. The total score is less than 13.
The change of Schirmer test | 1 week
  Standard tear test paper was taken and held in the conjunctival sac at 1/3 of the lower eyelid, and the patient was instructed to close the eyes gently. The results were observed 5 minutes later. Schirmer test < 10mm/5min was abnormal.

SECONDARY OUTCOMES:
Tear break-up time | 1 week
  After staining with 0.25% fluorescein sodium, patients were instructed to close their eyes under the slit lamp microscope. The tear film rupture time was calculated from the time of eye opening to the appearance of the first burst spot, and the mean value was taken for three consecutive tests. The tear film rupture time < 10s is abnormal
Fluorescein sodium staining of the ocular surface. | 1 week
  After staining with 0.25% fluorescein sodium, defect staining was observed under slit lamp microscope. Cornea was scored in 3 areas (FIG. 1) : top, center and bottom. Each area was scored according to 0 points (without any staining), 1 points (partial staining), 2 points (staining of more than half of the area) and 3 points (staining of the whole area), and the total was divided into the sum of 3 areas. A higher score indicates more severe ocular surface damage.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dana R, Bradley JL, Guerin A, Pivneva I, Stillman IO, Evans AM, Schaumberg DA. Estimated Prevalence and Incidence of Dry Eye Disease Based on Coding Analysis of a Large, All-age United States Health Care System. Am J Ophthalmol. 2019 Jun;202:47-54. doi: 10.1016/j.ajo.2019.01.026. Epub 2019 Feb 2. PMID 30721689
- [Result] Stapleton F, Alves M, Bunya VY, Jalbert I, Lekhanont K, Malet F, Na KS, Schaumberg D, Uchino M, Vehof J, Viso E, Vitale S, Jones L. TFOS DEWS II Epidemiology Report. Ocul Surf. 2017 Jul;15(3):334-365. doi: 10.1016/j.jtos.2017.05.003. Epub 2017 Jul 20. PMID 28736337
- [Result] Pflugfelder SC, de Paiva CS. The Pathophysiology of Dry Eye Disease: What We Know and Future Directions for Research. Ophthalmology. 2017 Nov;124(11S):S4-S13. doi: 10.1016/j.ophtha.2017.07.010. PMID 29055361
- [Result] Oguz H. Ocular surface disease and quality of life in patients with glaucoma. Am J Ophthalmol. 2012 May;153(5):1003; author reply 1003-4. doi: 10.1016/j.ajo.2012.01.017. No abstract available. PMID 22516154
- [Result] Baudouin C. Detrimental effect of preservatives in eyedrops: implications for the treatment of glaucoma. Acta Ophthalmol. 2008 Nov;86(7):716-26. doi: 10.1111/j.1755-3768.2008.01250.x. Epub 2008 Jun 3. PMID 18537937
- [Result] Yamaguchi T. Inflammatory Response in Dry Eye. Invest Ophthalmol Vis Sci. 2018 Nov 1;59(14):DES192-DES199. doi: 10.1167/iovs.17-23651. PMID 30481826
- [Result] Luo L, Li DQ, Doshi A, Farley W, Corrales RM, Pflugfelder SC. Experimental dry eye stimulates production of inflammatory cytokines and MMP-9 and activates MAPK signaling pathways on the ocular surface. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4293-301. doi: 10.1167/iovs.03-1145. PMID 15557435
- [Result] Fan NW, Dohlman TH, Foulsham W, McSoley M, Singh RB, Chen Y, Dana R. The role of Th17 immunity in chronic ocular surface disorders. Ocul Surf. 2021 Jan;19:157-168. doi: 10.1016/j.jtos.2020.05.009. Epub 2020 May 26. PMID 32470612
- [Result] Dohlman TH, Chauhan SK, Kodati S, Hua J, Chen Y, Omoto M, Sadrai Z, Dana R. The CCR6/CCL20 axis mediates Th17 cell migration to the ocular surface in dry eye disease. Invest Ophthalmol Vis Sci. 2013 Jun 12;54(6):4081-91. doi: 10.1167/iovs.12-11216. PMID 23702781
- [Result] De Paiva CS, Chotikavanich S, Pangelinan SB, Pitcher JD 3rd, Fang B, Zheng X, Ma P, Farley WJ, Siemasko KF, Niederkorn JY, Stern ME, Li DQ, Pflugfelder SC. IL-17 disrupts corneal barrier following desiccating stress. Mucosal Immunol. 2009 May;2(3):243-53. doi: 10.1038/mi.2009.5. Epub 2009 Feb 25. PMID 19242409
- [Result] Subbarayal B, Chauhan SK, Di Zazzo A, Dana R. IL-17 Augments B Cell Activation in Ocular Surface Autoimmunity. J Immunol. 2016 Nov 1;197(9):3464-3470. doi: 10.4049/jimmunol.1502641. Epub 2016 Sep 21. PMID 27655846
- [Result] Melnikov S, Mayan H, Uchida S, Holtzman EJ, Farfel Z. Cyclosporine metabolic side effects: association with the WNK4 system. Eur J Clin Invest. 2011 Oct;41(10):1113-20. doi: 10.1111/j.1365-2362.2011.02517.x. Epub 2011 Mar 24. PMID 21434893
- [Result] Park B, Lee IS, Hyun SW, Jo K, Lee TG, Kim JS, Kim CS. The Protective Effect of Polygonum cuspidatum (PCE) Aqueous Extract in a Dry Eye Model. Nutrients. 2018 Oct 19;10(10):1550. doi: 10.3390/nu10101550. PMID 30347752
- [Result] Perry HD, Solomon R, Donnenfeld ED, Perry AR, Wittpenn JR, Greenman HE, Savage HE. Evaluation of topical cyclosporine for the treatment of dry eye disease. Arch Ophthalmol. 2008 Aug;126(8):1046-50. doi: 10.1001/archopht.126.8.1046. PMID 18695097
- [Result] de Paiva CS, Pflugfelder SC, Ng SM, Akpek EK. Topical cyclosporine A therapy for dry eye syndrome. Cochrane Database Syst Rev. 2019 Sep 13;9(9):CD010051. doi: 10.1002/14651858.CD010051.pub2. PMID 31517988
- [Result] Holland EJ, Darvish M, Nichols KK, Jones L, Karpecki PM. Efficacy of topical ophthalmic drugs in the treatment of dry eye disease: A systematic literature review. Ocul Surf. 2019 Jul;17(3):412-423. doi: 10.1016/j.jtos.2019.02.012. Epub 2019 Mar 4. PMID 30844466
- [Result] Prockop DJ, Kota DJ, Bazhanov N, Reger RL. Evolving paradigms for repair of tissues by adult stem/progenitor cells (MSCs). J Cell Mol Med. 2010 Sep;14(9):2190-9. doi: 10.1111/j.1582-4934.2010.01151.x. PMID 20716123
- [Result] Han Y, Yang J, Fang J, Zhou Y, Candi E, Wang J, Hua D, Shao C, Shi Y. The secretion profile of mesenchymal stem cells and potential applications in treating human diseases. Signal Transduct Target Ther. 2022 Mar 21;7(1):92. doi: 10.1038/s41392-022-00932-0. PMID 35314676
- [Result] Prockop DJ, Oh JY. Mesenchymal stem/stromal cells (MSCs): role as guardians of inflammation. Mol Ther. 2012 Jan;20(1):14-20. doi: 10.1038/mt.2011.211. Epub 2011 Oct 18. PMID 22008910
- [Result] Yao G, Qi J, Liang J, Shi B, Chen W, Li W, Tang X, Wang D, Lu L, Chen W, Shi S, Hou Y, Sun L. Mesenchymal stem cell transplantation alleviates experimental Sjogren's syndrome through IFN-beta/IL-27 signaling axis. Theranostics. 2019 Oct 21;9(26):8253-8265. doi: 10.7150/thno.37351. eCollection 2019. PMID 31754394
- [Result] Li Y, Ma K, Zhang L, Xu H, Zhang N. Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells Alleviate Dextran Sulfate Sodium-Induced Colitis by Increasing Regulatory T Cells in Mice. Front Cell Dev Biol. 2020 Nov 24;8:604021. doi: 10.3389/fcell.2020.604021. eCollection 2020. PMID 33330503
- [Result] Lee MJ, Ko AY, Ko JH, Lee HJ, Kim MK, Wee WR, Khwarg SI, Oh JY. Mesenchymal stem/stromal cells protect the ocular surface by suppressing inflammation in an experimental dry eye. Mol Ther. 2015 Jan;23(1):139-46. doi: 10.1038/mt.2014.159. Epub 2014 Aug 25. PMID 25152016
- [Result] Villatoro AJ, Fernandez V, Claros S, Rico-Llanos GA, Becerra J, Andrades JA. Use of adipose-derived mesenchymal stem cells in keratoconjunctivitis sicca in a canine model. Biomed Res Int. 2015;2015:527926. doi: 10.1155/2015/527926. Epub 2015 Feb 23. PMID 25802852
- [Result] Sgrignoli MR, Silva DA, Nascimento FF, Sgrignoli DAM, Nai GA, da Silva MG, de Barros MA, Bittencourt MKW, de Morais BP, Dinallo HR, Foglia BTD, Cabrera WB, Fares EC, Andrade SF. Reduction in the inflammatory markers CD4, IL-1, IL-6 and TNFalpha in dogs with keratoconjunctivitis sicca treated topically with mesenchymal stem cells. Stem Cell Res. 2019 Aug;39:101525. doi: 10.1016/j.scr.2019.101525. Epub 2019 Jul 31. PMID 31430719
- [Derived] Zhang D, Chen T, Liang Q, Feng X, Jiang J, Chen Z, Tang Y, Chu Y, Wang B, Hu K. A first-in-human, prospective pilot trial of umbilical cord-derived mesenchymal stem cell eye drops therapy for patients with refractory non-Sjogren's and Sjogren's syndrome dry eye disease. Stem Cell Res Ther. 2025 Apr 23;16(1):202. doi: 10.1186/s13287-025-04292-8. PMID 40269970